CLINICAL TRIAL: NCT01538992
Title: Phase 3 Study of Renal Denervation That Improves Symptoms of Heart Failure and Enhances Life Quality in Advanced Heart Failure
Brief Title: Renal Denervation in Patients With Advanced Heart Failure
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: we could not fined enough patients for the study
Sponsor: Bursa Postgraduate Hospital (Other)
Responsible Party: Principal Investigator, Hasan ARI, Medical Doctor, Cardiology Chief Intern, Bursa Postgraduate Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bursa YİEAH
Record Dates: First submitted 2012-02-16; First posted 2012-02-27 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Heart Failure
Keywords: renal denervation; heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- renal denervation (Experimental): in this group percutaneous renal denervation with Standard steerable Mariner Radiofreqency ablation Catheter (5F or 7F)
  Interventions: Device: Standard steerable Marinr RF ablation Catheter (5F or 7F)
- medical thrapy (No Intervention): medical treatment

INTERVENTIONS:
Device: Standard steerable Marinr RF ablation Catheter (5F or 7F) — Intervention: Device: Standard steerable Mariner Radiofrequency ablation Catheter (5F or 7F)
  Other Names: Renal ablation
  Arms: renal denervation

SUMMARY:
Sympathetic system has important role occurrence of symptoms in heart failure. Renal denervation that is ablated some of sympathetic nerves is affected pathology of heart failure. This interventional therapy improves symptoms and life quality.

DETAILED DESCRIPTION:
Primary Outcome Measures:

• Safety of Renal Denervation in Heart Failure patients as measured by Adverse Events

Secondary Outcome Measures:

• Ventricular function,NYHA functional Class, 6 min walking test, biochemical test and Renal function as measured by Glomerular Filtration Rate (GFR)

Eligibility Patients population: Volunteers, NYHA Class III-IV heart failure patients. Ages Eligible for Study: 18 Years to 85 Years Genders Eligible for Study: Both Accepts Healthy Volunteers: No

ELIGIBILITY:
Inclusion Criteria:

* Heart Failure patients NYHA Class III or IV
* Left Ventricular Ejection Function < 35%
* GFR > 45 mL/min/1.73m2
* Optimal stable medical therapy

Exclusion Criteria:

* Do not eligible renal artery anatomy for treatment as determined by Angiography, and
* History of prior renal artery intervention
* Single functioning kidney.
* Myocardial Infarction, unstable angina pectoris or cerebrovascular Accident within 3 months
* Systolic BP < 110mmHG Hospitalisation because of heart failure in last 3 weeks.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2014-01 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Safety of Renal Denervation in Heart Failure patients as measured by Adverse Events | 6 months

SECONDARY OUTCOMES:
• Ventricular function as measured by Echocardiography • NYHA functional Class, 6 min walking test, biochemical test. • Renal function as measured by Glomerular Filtration Rate (GFR) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: HASAN ARI, MD, Study Director — Bursa Postgraduate Hospital
Locations (1):
- Bursa Yüksek İhtisas Eğitim ve Araştırma Hastanesi, Bursa, Turkey (Türkiye)